CLINICAL TRIAL: NCT04352270
Title: A Randomized Controlled Study of Clinic-Based Atopic Dermatitis Therapeutic Patient Education
Brief Title: Clinic-Based Atopic Dermatitis Therapeutic Patient Education
Acronym: AD-TPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-39538
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
Keywords: Therapeutic patient education; Printed handouts; Educational videos; Child-parent dyads
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Printed educational materials (Active Comparator): Parent-child dyads randomized to this group will receive printed educational materials in English or Spanish about atopic dermatitis.
  Interventions: Other: AD printed educational materials
- Group 2- Educational videos (Experimental): Parent-child dyads randomized to this group will receive an investigator developed educational video in English or Spanish about atopic dermatitis.
  Interventions: Other: AD educational videos

INTERVENTIONS:
Other: AD printed educational materials — Printed educational materials in Spanish and English about coping with Atopic Dermatitis, specifically geared towards children and parents will be given to participants.
  Arms: Group 1- Printed educational materials
Other: AD educational videos — Short, educational videos in English and Spanish about coping with Atopic Dermatitis, specifically geared towards children and parents will be developed. There will be Spanish and English versions of the videos, minimal text, comprehensive language, animations, and it will be administered via user friendly platforms or websites.
  Arms: Group 2- Educational videos

SUMMARY:
The primary objective of this randomized trial is to determine whether comprehensive, accessible, and animation-style videos are a more effective method of therapeutic patient education (TPE) based on clinical outcomes than paper handouts in Spanish and English-speaking communities. The clinical outcomes being measured are the severity, sleep affected by atopic dermatitis (AD), and the amount of itch experienced.

DETAILED DESCRIPTION:
Patients will be recruited, stratified, and then randomly assigned into one of two intervention groups.The patient participants will be children anywhere on the spectrum of mild to severe AD and they will be stratified into four strata: a) Those with severe AD and no medical intervention escalation, b) Those with mild AD and no medical intervention escalation, c) Those with severe AD and medical intervention escalation, and d) Those with mild AD and medical intervention escalation. Group 1 will be a paper handout for group 1 and an educational video for group 2 as a form of TPE. Subjects will be recruited in clinic after they are screened for AD during their regular dermatology appointment. The research team will provide the patient and parent with a brief introduction to the study, what it involves for the patient, any foreseeable risks, and the compensation. If they agree to participate, a consent/permission form will be given to the parent/guardian to sign. After an initial evaluation of the patient's AD, subjects will receive an initial survey and POEM questionnaire on an iPad via RedCap that will address the condition of their AD. The patient will be administered a form of TPE as the intervention. The intervention will first be viewed/read in clinic, followed by a brief set of questions from the research team to determine the amount of information retained on an immediate level. A follow-up appointment will be scheduled for the patient. Group 2 will receive a slip of paper with a link to the videos, so the TPE will be accessible outside the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Boston Medical Center (BMC) patients under the age of 18 diagnosed with AD and their parents/legal guardian
* Spanish or English speakers
* Have access to the internet

Exclusion Criteria:

* None

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Change in eczema severity based on the Patient Oriented Eczema Measure (POEM) | baseline, up to 2 months
  The Patient Oriented Eczema Measure (POEM) is a validated 7 item instrument with response categories from 0 to 4 where No days = 0, 1-2 days = 1, 3-4 days = 2, 5-6 days = 3, Every day = 4. Scoring for the POEM ranges form 0 to 28 and is interpreted by 0 to 2 = Clear or almost clear, 3 to 7 = Mild eczema, 8 to 16 = Moderate eczema, 17 to 24 = Severe eczema, 25 to 28 = Very severe eczema.
Change in eczema severity based on the Eczema Area and Severity Index (EASI) | baseline, up to 2 months
  The Eczema Area and Severity Index (EASI) is an investigator-assessed instrument measuring the severity of clinical signs in atopic dermatitis (AD). The suggested severity strata for the EASI are: 0 = clear; 0·1-1·0 = almost clear; 1·1-7·0 = mild; 7·1-21·0 = moderate; 21·1-50·0 = severe; 50·1-72·0 = very severe
Change in the severity of itch | baseline, up to 2 months
  An investigator developed survey completed by participants with questions about itch will be used to collect data to assess this outcome.
Change in sleep quality | baseline, up to 2 months
  An investigator developed survey completed by participants with questions about sleep quality will be used to collect data to assess this outcome.

SECONDARY OUTCOMES:
Change in the overall quality of life | baseline, up to 2 months
  An investigator developed survey completed by participants with questions about quality of life will be used to collect data to assess this outcome.
Change in patient/parent confidence | baseline, up to 2 months
  An investigator developed survey completed by participants with questions about confidence will be used to collect data to assess this outcome.
Change in knowledge of coping with Atopic Dermatitis (AD) | baseline, up to 2 months
  An investigator developed survey completed by participants with questions about their knowledge of coping with AD will be used to collect data to assess this outcome.
Satisfaction with therapeutic patient education (TPE) | up to 2 months
  An investigator developed survey completed by participants with questions about their satisfaction about TPE will be used to collect data to assess this outcome.
Atopic Dermatitis related costs | 6 months
  Billing records will be analyzed to assess AD related costs.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lee, MD PhD, Principal Investigator — Boston University
Locations (1):
- BMC Pediatric Dermatology Clinics, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No